CLINICAL TRIAL: NCT05038852
Title: Acceptability of Mobile Applications (Apps) to Enhance Smoking Cessation in a Clinical Tobacco Treatment Program - A Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0984; NCI-2021-09413 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-08-25; First posted 2021-09-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Tobacco
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 smartphone applications (Other): app is designed to help you learn relaxation skills
  Interventions: Device: smartphone applications
- Group 2 smartphone applications (Other): app is designed to help you increase your positive feelings, behaviors, and thoughts.
  Interventions: Device: smartphone applications

INTERVENTIONS:
Device: smartphone applications — app is designed to help you learn relaxation skills.
Device: smartphone applications — app is designed to help you increase your positive feelings, behaviors, and thoughts.

SUMMARY:
We will conduct a small-scale randomized controlled trial (RCT) with 24 adult smokers enrolled in the TTP. Participants will receive either the Free4Good mobile app for positive psychology skills training or a breathing relaxation mobile app control (Breathe2Relax). All participants will be receiving tobacco cessation treatment in the Tobacco Treatment Program at MD Anderson as standard of care.

DETAILED DESCRIPTION:
The aims of this pilot protocol are to test the adherence, acceptability, user satisfaction, and preliminary efficacy of a smartphone mobile health app, Free4Good, which incorporates skills training in positive psychology vs. a relaxation app, Breathe2Relax (control condition), in a small randomized controlled trial of smokers (N = 24). Adherence will be measured directly through app usage data. Acceptability and user satisfaction will be measured via specific items included on a User Satisfaction Questionnaire. Efficacy outcomes include evidence of increased engagement in positive psychology-related quitting strategies (measured by the Quitting Strategies Questionnaire) and smoking abstinence.

Exploratory analyses including covariates such as nicotine dependence, mood, and depressive symptoms may be examined as appropriate, as these measures have been shown to predict abstinence outcomes in a variety of studies.1-4 Changes in mood and/or depressive symptoms may also be characterized

ELIGIBILITY:
Inclusion criteria:

* MD Anderson patient between the ages of 18 to 65
* current smoker (i.e., at least 1 cigarette or e-cig per day)
* smoking for at least one year,
* willing to set a quit date in the next 30 days,
* not engaged in smoking cessation treatment other than the MDACC Tobacco Treatment Program
* English speaking and ability to read and comprehend English, and 7) currently own an iOS mobile phone (iPhone) using iOS 9.0 or later and reports regular use (at least weekly) of at least 1 iOS app.

Exclusion Criteria

* endorsing current suicidal ideation or intent,
* meeting criteria for a current Major Depressive Episode measured by the PHQ-9,
* any medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator or Collaborator,
* subject considered by the investigator an unsuitable candidate for receipt of a smoking cessation treatment or unstable to be followed up throughout the entire duration of the study.
* Pregnant women will not be excluded from participating in the study and any decisions about potential pharmacotherapy will be done as standard of care in the Tobacco Treatment Program, including a consultation with the medical team and a joint decision-making process with the patient to determine the best course of treatment given all co-morbid medical conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To assess the adherence of a smartphone mobile health app. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Minnix, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org